CLINICAL TRIAL: NCT02460328
Title: Resolution of Primary Immune Defect in 22q11.2 Deletion Syndrome
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 794/2557(EC4)
Record Dates: First submitted 2015-04-10; First posted 2015-06-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Immune Defect; 22q11.2 Deletion Syndrome
MeSH Terms: conditions — DiGeorge Syndrome

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
* Evaluate about age of resolution in immune defect in 22q11.2 Deletion Syndrome
* Incidence of immunodeficiencies in 22q11.2 Deletion Syndrome

DETAILED DESCRIPTION:
22q11.2 Deletion Syndrome is the most common for microdeletion syndrome. The incidence is about 1:4000 of live birth. Clinical features in this syndrome are vary which consist of conotruncal cardiac anomalies, developmental disabilities, palatal anomalies, speech delay, hypocalcemia, characteristic facial features and immunodeficiencies. The most common type of immunodeficiencies is T cell defect that associated with thymic hypoplasia. In the present time, the investigators don't know about the resolution of immune defect in this syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 22q11.2 deletion syndrome patients in allergy and immunology clinic, genetic clinic, cardio clinic, genetic clinic and development clinic

Exclusion Criteria:

* loss follow up in 22q11.2 deletion syndrome patients or incomplete medical record

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 22q11.2 deletion syndrome diagnosed from Fluorescence in situ hybridization (FISH) for 22q11
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
age of resolution in immune defect in 22q11.2 Deletion Syndrome | 18 months

SECONDARY OUTCOMES:
incidence of immunodeficiencies in 22q11.2 Deletion Syndrome | 18 months
type of infectious disease in 22q11.2 Deletion Syndrome | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD., Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] McLean-Tooke A, Barge D, Spickett GP, Gennery AR. Immunologic defects in 22q11.2 deletion syndrome. J Allergy Clin Immunol. 2008 Aug;122(2):362-7, 367.e1-4. doi: 10.1016/j.jaci.2008.03.033. Epub 2008 May 16. PMID 18485468
- [Result] Chinen J, Rosenblatt HM, Smith EO, Shearer WT, Noroski LM. Long-term assessment of T-cell populations in DiGeorge syndrome. J Allergy Clin Immunol. 2003 Mar;111(3):573-9. doi: 10.1067/mai.2003.165. PMID 12642839